CLINICAL TRIAL: NCT03344718
Title: Inverse Relationship Between Metabolic Syndrome and Vitamin D Level in Old People Without Vitamin D Deficiency
Brief Title: Metabolic Syndrome and Vitamin D Level in Old People
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hsing Wu, Associate Professor, National Cheng-Kung University Hospital
Other Study IDs: Tianliao old people study 2012
Record Dates: First submitted 2017-09-10; First posted 2017-11-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2017-11

CONDITIONS: Elderly; Metabolic Syndrome; Vitamin D Deficiency; Ostreocalcin; Insulin Resistance; Obesity; Osteoporosis; Sarcopenia
MeSH Terms: conditions — Metabolic Syndrome; Vitamin D Deficiency; Insulin Resistance; Obesity; Osteoporosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples Without DNA — Centrifuged blood serum (5 ml) was stored in -80'C refrigerator for each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2012, a cross-sectional survey sampling 1,966 community-dwelling old people was conducted. Structurized questionnaires were interviewed face-to-face by well-trained staffs. An overnight fasting blood were obtained for biochemistry parameters.

ELIGIBILITY:
Inclusion Criteria:

* more than 65-year-old

Exclusion Criteria:

* excluding empty houses, death, non-ambulatory subjects (subjects with significant disabilities, such as handicapped cerebral vascular accident, cancerous cachexia, unstable chronic diseases or psychiatric disorders, severe arthritis or inflammatory disease), uncomfortable anorexia by any medications, and non-reachable subjects

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Tianliao District, located in Kaohsiung City in southern Taiwan, is a tropical, agriculture-based community. It is located at around 22N50' latitude, like Hawaii (18° 55' N to 28° 27' N), and about 7° farther south than Florida (24° 27' N to 31° 00' N). The annual average temperature is 25.1°C (range: 19.3-29.2°C), and its annual average sunshine duration is 212.2 hours (longest: 221.4 hours in July; shortest: 161.8 hours in December). In the 2012 census report, the total population of Tianliao District was 7800, and 1966 (25.2%) participants were ≥ 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2012-08-17 (Actual); Study Completion 2012-08-17 (Actual)

PRIMARY OUTCOMES:
Osteoporotic fracture rate | 5 year
  Vertebra, non-vertebra, major fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Family Medicine, National Cheng Kung Univ Hosp, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CH, Chen KT, Hou MT, Chang YF, Chang CS, Liu PY, Wu SJ, Chiu CJ, Jou IM, Chen CY. Prevalence and associated factors of sarcopenia and severe sarcopenia in older Taiwanese living in rural community: the Tianliao Old People study 04. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:69-75. doi: 10.1111/ggi.12233. PMID 24450563